CLINICAL TRIAL: NCT01257529
Title: An Open-Label, Single-Dose, Randomized, Four-Way Crossover Study In Healthy Volunteers To Evaluate The Effects Of A Low, Medium And High Fat Evening Meal On The Pharmacokinetics Of Pregabalin Controlled Release Formulation As Compared To The Immediate Release Formulation
Brief Title: An Investigation Of The Absorption And Pharmacokinetics Of A Single Dose Of A Controlled Release (CR) Pregabalin Tablet Following A Low, Medium, And High-Fat Evening Meal As Compared To A Single Dose Of The Immediate Release (IR) Pregabalin Capsule In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081227
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability; bioequivalence
MeSH Terms: interventions — Diet, Fat-Restricted; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin controlled release, 330 mg, low-fat (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, low-fat
- Pregabalin controlled release, 330 mg, medium-fat (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, medium-fat
- Pregabalin controlled release, 330 mg, high-fat (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, high-fat
- Pregabalin immediate release, 300 mg (Other): Reference Treatment
  Interventions: Drug: Pregabalin immediate release, 300 mg

INTERVENTIONS:
Drug: Pregabalin controlled release, 330 mg, low-fat — A single oral dose of 330 mg controlled release tablet administered following a low-fat evening meal
  Arms: Pregabalin controlled release, 330 mg, low-fat
Drug: Pregabalin controlled release, 330 mg, medium-fat — A single oral dose of 330 mg controlled release tablet administered following a medium-fat evening meal
  Arms: Pregabalin controlled release, 330 mg, medium-fat
Drug: Pregabalin controlled release, 330 mg, high-fat — A single oral dose of 330 mg controlled release tablet administered following a high-fat evening meal
  Arms: Pregabalin controlled release, 330 mg, high-fat
Drug: Pregabalin immediate release, 300 mg — A single oral dose of 300 mg immediate release capsule administered following a medium-fat evening meal
  Arms: Pregabalin immediate release, 300 mg

SUMMARY:
The purpose of this study is to 1) evaluate the extent of absorption of a single dose of a pregabalin controlled release tablet following either a low, medium, or high-fat evening meal as compared to a single dose of the pregabalin immediate release capsule, 2) evaluate the safety and tolerability of a single dose of a pregabalin controlled release tablet following a low, medium, or high fat evening meal as compared to a single dose of the pregabalin immediate release capsule.

DETAILED DESCRIPTION:
Evaluate the absorption, pharmacokinetics, safety/tolerability of a single dose of a pregabalin CR tablet under various conditions as compared to single dose of pregabalin IR capsule

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve from 0 to infinity (AUCinf) for assessment of equivalence between the controlled release treatments and the immediate release treatments | 3 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Chew ML, Plotka A, Alvey CW, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pharmacokinetics of pregabalin controlled-release in healthy volunteers: effect of food in five single-dose, randomized, clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):617-26. doi: 10.1007/s40261-014-0211-4. PMID 25078976
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081227